CLINICAL TRIAL: NCT04767230
Title: The Effect of a Healthy Diet Containing Flaxseed and Olive Oil Compared With Healthy Dietary Advice on Cardiovascular Disease Risk Markers in Patients With Coronary Artery Disease
Brief Title: The Effect of a Healthy Diet Containing Flaxseed and Olive Oil on Cardiovascular Disease Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nafiseh Khandouzi, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25672
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A heart-healthy diet + Flaxseed + Olive oil (Active Comparator): A heart-healthy diet with a specified number of food servings from different food groups (including vegetables, fruits, grains, dairy products, meats) + daily consumption of 30 grams of flaxseed + 25 mL/day of refined olive oil (equivalent to 4 tablespoons; 2 tablespoons for lunch and 2 tablespoons for dinner) for 3 months
  Interventions: Other: Dietary Intervention
- A heart-healthy diet (Placebo Comparator): Recommendations for a heart-healthy diet, such as those of the American Heart Association for 3 months. These include eating at least 5 servings of vegetables and fruits daily, reduction in the consumption of sources of saturated and trans fats by avoiding the consumption of high-fat red meats and replacing them with low-fat meat or with poultry and fish, replacing low-fat dairy sources with regular or high-fat ones; consumption of regular vegetable oils such as canola and sunflower; reduction in salt consumption; and reduction in the consumption of simple sugars for 3 months
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — A heart-healthy diet + daily consumption of 30 grams of flaxseed + 25 mL/day of refined olive oil in adjunct to medical treatment for 3 months

SUMMARY:
Flaxseed and olive oil consumption have beneficial effects on cardiovascular risk factors. Nonetheless the effects of their simultaneous consumption have not yet been studied.The purpose of this study is to investigate the effects of a healthy diet containing flaxseed and olive oil compared with healthy dietary advice on cardiovascular disease risk markers in patients with coronary artery disease (CAD), in improving flow-mediated dilation, plasma lipid profile and fatty acids composition of red blood cells.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be conducted in Rajaie Cardiovascular Center in Tehran, Iran. After review of the inclusion and exclusion criteria and explanation of the design of the study, written consent form will be completed. The participants are 50 eligible coronary artery disease patients, aged 30-75 years. Intervention group will be received a heart-healthy diet with a specified number of food servings from different food groups (including vegetables, fruits, grains, dairy products, meats) + daily consumption of 30 grams of flaxseed + 25 mL/day of refined olive oil (equivalent to 4 tablespoons; 2 tablespoons for lunch and 2 tablespoons for dinner); and control group will be received recommendations for a heart-healthy diet, such as those of the American Heart Association for 3 months. These include eating at least 5 servings of vegetables and fruits daily, reduction in the consumption of sources of saturated and trans fats by avoiding the consumption of high-fat red meats and replacing them with low-fat meat or with poultry and fish, replacing low-fat dairy sources with regular or high-fat ones; consumption of regular vegetable oils such as canola and sunflower; reduction in salt consumption; and reduction in the consumption of simple sugars, for 3 months. Flow mediated dilatation (FMD) in brachial artery via ultrasonography, plasma levels of lipids and lipoproteins via enzymatic method, and fatty acids composition of red blood cells via gas chromatography method were measured.

ELIGIBILITY:
Inclusion Criteria:

1. Established coronary artery disease as verified by coronary angiography
2. Body ass index <30 kg/m2
3. men and postmenopausal women
4. Willing to participate in the study

Exclusion Criteria:

1. Unwilling to follow the protocol and/or give informed consent
2. Chronic Kidney Disease stage 4 or 5 or a reported history cancer
3. Regular consumption of flaxseed or omega-3 supplements during previous month
4. Any changes in the disease treatment plan including type or dose of lipid-lowering medications or coronary artery bypass graft during the study period

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Flow Mediated Dilation (FMD) in brachial artery | 3 months
  Measurement of dilation of the brachial artery by ultrasonography from baseline to 3 months later

SECONDARY OUTCOMES:
Plasma lipid profile (total cholesterol, LDL-C, HDL-C, triglyceride) | 3 months
  Measurement of plasma level of lipid profile by enzymatic method from baseline to 3 months later
Total fatty acids composition of red blood cells | 3 months
  Measurement of total fatty acids composition of red blood cells by gas chromatography from baseline to 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nasrollahzadeh, Ph.D, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edel AL, Rodriguez-Leyva D, Maddaford TG, Caligiuri SP, Austria JA, Weighell W, Guzman R, Aliani M, Pierce GN. Dietary flaxseed independently lowers circulating cholesterol and lowers it beyond the effects of cholesterol-lowering medications alone in patients with peripheral artery disease. J Nutr. 2015 Apr;145(4):749-57. doi: 10.3945/jn.114.204594. Epub 2015 Feb 18. PMID 25694068
- [Background] Khandouzi N, Zahedmehr A, Mohammadzadeh A, Sanati HR, Nasrollahzadeh J. Effect of flaxseed consumption on flow-mediated dilation and inflammatory biomarkers in patients with coronary artery disease: a randomized controlled trial. Eur J Clin Nutr. 2019 Feb;73(2):258-265. doi: 10.1038/s41430-018-0268-x. Epub 2018 Aug 20. PMID 30127374
- [Background] Mandasescu S, Mocanu V, Dascalita AM, Haliga R, Nestian I, Stitt PA, Luca V. Flaxseed supplementation in hyperlipidemic patients. Rev Med Chir Soc Med Nat Iasi. 2005 Jul-Sep;109(3):502-6. PMID 16607740
- [Background] Bloedon LT, Balikai S, Chittams J, Cunnane SC, Berlin JA, Rader DJ, Szapary PO. Flaxseed and cardiovascular risk factors: results from a double blind, randomized, controlled clinical trial. J Am Coll Nutr. 2008 Feb;27(1):65-74. doi: 10.1080/07315724.2008.10719676. PMID 18460483